CLINICAL TRIAL: NCT06777849
Title: Mainstreaming a Life Skills Education Programme Right to Play- Plus to Reduce Violence Against Girls in Pakistan
Acronym: RTP-Plus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: George Washington University (Other)
Responsible Party: Principal Investigator, Dr Rozina Karmaliani, Professor & Associate Director, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-9681-30134; 22-SC35-INT (Other: The George Washington University)
Record Dates: First submitted 2025-01-02; First posted 2025-01-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Mental Health; Gender Based Violence; Resilience; Gender Equity; Sexual and Reproductive Health and Rights
Keywords: GBV; adolescent health; play-based life skills; what works
MeSH Terms: conditions — Psychological Well-Being; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention arm participants will receive the adapted play-based life skills education intervention from teachers, which the Right to Play and Aahung will deliver.
  Interventions: Behavioral: Right to Play-Plus (RTP-Plus)
- Control (Other): The control arm will not receive the intervention during the two years of cluster randomised control trial (cRCT). However, a delayed intervention will be offered to the control arm upon completion of endline data collection after the comprehensive intervention is delivered in the intervention arm.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Right to Play-Plus (RTP-Plus) — The comprehensive curriculum comprises of themes: "Social and Emotional Development" and "Sexual and Reproductive Health" will be delivered by school teachers who will receive training from Right to Play and Aahung. There will be 60 sessions for two years.
  Other Names: What Works 2
  Arms: Intervention
Other: Control — There will be no intervention given to control arm during two years of cluster randomised control trial (cRCT). However, a delayed intervention having teachers' training, will be provided to the control arm after the completion of endline for the duration of 3-4 months.
  Arms: Control

SUMMARY:
Right to Play-Plus (RTP-Plus) aims to address violence against women and girls by promoting changes in social norms among young people within the school environment. The project focuses on building the capacity of young people to identify harmful gender norms and prevent violence against girls and boys by incorporating Right to Play's play-based learning methodology and Aahung's Life Skills Based Education curriculum. The strategies employed include interactive, learner-centered methodologies, curricular activities, and the development of peer educators and junior leaders. Teachers play a crucial role as key influencers and delivery agents of the curricular content. The project emphasizes capacity development for teachers, challenging their social norms, strengthening their play-based methodologies, and improving their sexual and reproductive health and rights knowledge (SRHR). The ultimate goal is to equip teachers to effectively deliver a gender transformative curriculum, empowering young people to respond to and prevent violence.

The research question for this study is:

What is the effectiveness of an adapted play-based life skills education that incorporates a "whole school" approach in reducing sexual harassment and abuse, peer violence experiences, mental illness (including suicidal ideation), improving resilience, and promoting gender equity, SRHR knowledge in both home and public settings?

The research objective will be achieved through two-arm cluster randomized controlled trial (for girls-only, co-ed, and boys-only schools). The intervention arm participants will be able to participate in the adapted play-based life skills education intervention, which the Right to Play and Aahung will deliver. It will be provided to all eligible school children in grade 6. Moreover, a delayed intervention will be offered to the control arm upon completion of endline data collection after the comprehensive intervention is delivered in the intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* Schools will be chosen from District Malir and adjacent areas, including Korangi and East Karachi. Among the 100 selected schools, the following distribution will be maintained: 40 girls-only schools (public), 40 co-ed schools (private), and 20 boys-only schools (public).
* Schools having a minimum of 30 students enrolled in grade 6
* Private schools with low to medium fees, with monthly amounts ranging from PKR 2000 to 3500.
* Factors such as teacher availability, school management support, accessibility to research and intervention partners, and school clustering will also be considered for the selection of these hundred schools.
* Schools' willingness to adapt child protection and safeguarding/anti-harassment administrative measures and policies to improve school safety, reduce the use of corporal punishment, enhance school performance, and increase girls' retention rates, primarily apply to private schools.

Exclusion Criteria:

* Schools where Right to Play or Aahung have already implemented their play-based/other activities.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in physical, emotional, and sexual violence | From enrollment to the end of intervention after 2 years.
  International Society for Prevention of Child Abuse and Neglect (ISPCAN)-Child Abuse Screening Tool for children (ICAST-C) is used to measure physical, emotional and sexual violence at home among children aged 11 to 18 years. It has been adapted for use in school settings in previous studies to measure child abuse at school. 12 items related to physical and emotional violence, and 9 items related to sexual violence will be used in the current study to measure physical, emotional and sexual violence at home, school, and community. Each item is measured if this incident happened with the child or not. If yes, then next column measures whether it happened in the past 4 weeks or not. Moreover, there are questions about the location of such an incident and the person who perpetrated it. These questions will yield data on the proportion of children affected by physical, emotional, and sexual violence, the location of perpetration, and the characteristics of perpetrators.
Change in cyber sexual harassment | From enrollment to the end of the intervention after 2 years.
  Following the same pattern of International Society for Prevention of Child Abuse and Neglect (ISPCAN)-Child Abuse Screening Tool for Children (ICAST-C) questions to measure physical, emotional, and sexual violence, a self-developed 6-item scale will be used to measure the prevalence (with answers yes (1), no (0), or don't know (-99)) of cyber sexual violence, its frequency in the past 4 weeks and the information on location and perpetrators. These questions will yield data on the proportion of children affected by cyber sexual violence, the location of perpetration, and the characteristics of perpetrators.
Increased self-efficacy to respond to violence | From enrollment to the end of intervention after 2 years.
  A self-developed 2-item scale adapted from the Self-Efficacy to Deal with Violence Scale to measure confidence in responding to an act of violence. All items will be measured on a binary scale from 0 to 1 where 0 (No) refers to not confident, and 1 (Yes) refers to confident. The results will reflect the proportion of having confidence in responding to violence.

SECONDARY OUTCOMES:
Change in attitudes towards gender equality | From enrollment to the end of intervention after 2 years.
  A 5-item scale was adapted from Nancy Perrin, et al (2019) to measure the personal beliefs of children about gender equality. All items will be measured on a binary scale from 0 to 1 where 0 refers to disagree, and 1 refers to agree. Item 1 will be reverse coded. The results will reflect the proportion of having progressive gender beliefs.
Change in acceptability of violence against women | From enrollment to the end of intervention after 2 years.
  An adapted scale from Nancy Perrin, et al (2019) will be used to measure personal beliefs of justifying a man to hit his wife. All 6 items will be measured on a binary scale from 0 to 1 where 0 (no) refers to disagree, and 1 (yes) refers to agree. The results will reflect the proportion of respondents with conservative beliefs accepting domestic violence against women.
Change in beliefs about child marriage | From enrollment to the end of intervention after 2 years.
  An adapted 5-item scale from Perrin, N et al, 2019 to measure personal beliefs about girls being married at an early age. All items will be measured on a binary scale from 0 to 1 where 0 refers to disagree, and 1 refers to agree. Item 5 will be reverse-coded. The overall score ranges from 0 to 5, with higher scores reflecting conservative beliefs accepting child marriage.
Change in peer violence perpetration | From enrollment to the end of intervention after 2 years.
  A 10-item scale adapted from the peer perpetration scale from the Multidimensional Scale of Peer Violence is used to measure physical and emotional violence. All items will be measured on a binary scale from 0 to 1 where 0 (No) refers to did not do the act, and 1 (Yes) refers to did the act. The overall score ranges from 0 to 10, with higher scores reflecting the carrying out of the act of peer perpetration violence.
Increased resilience | From enrollment to the end of intervention after 2 years.
  The 10-item Connor-Davidson Resilience Scale (CD-RISC-10) was extracted from the original 25-item Connor-Davidson Resilience Scale (CD-RISC-25)(Campbell-Sills and Stein, 2007). Item responses range from 0 ("not true at all") to 4 ("true nearly all of the time"). The overall score ranges from 0 to 40, with higher scores reflecting a greater ability to cope with adversity.
Change in depression | From enrollment to the end of intervention after 2 years.
  The Patient Health Questionnaire 9 will be used to measure depression. All items will be measured on a binary scale from 0 to 1 where 0 refers to Not at All, and 1 refers to Yes (at least once or more). The results will reflect the proportion of symptoms of depression.
Change in sexual health confidence | From enrollment to the end of intervention after 2 years.
  This is a secondary outcome that the intervention partners will observe. This will be assessed with a self-developed tool with 5 items. It comprises of 5-point Likert scale to rate the individual's evaluation ranging from 1 (Strongly Disagree) to 5 (Strongly Agree), where higher scores mean more confident.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Korangi, Karachi, Sindh
  - Malir, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No
The personal identification of participants will not be disclosed to anyone, and identifiers will not be included in the dataset. Data analysis will be done using unique codes assigned to participants per their categories. All research findings will be written up so the identity of participants will be concealed.